CLINICAL TRIAL: NCT05061823
Title: An Open-label, Multicenter Follow-up Study to Collect Long-term Data on Participants From Multiple Bintrafusp Alfa (M7824) Clinical Studies
Brief Title: Bintrafusp Alfa Program Rollover Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS200647_0054; 2021-000179-36 (EudraCT Number)
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Cancer
Keywords: Solid Tumors; Tumor response; Safety; Efficacy; Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST1.1); Programmed death ligand 1; Survival Follow-up; Human transforming growth factor β (TGFβ) receptor II; Performance Status; Bintrafusp alfa
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bintrafusp alfa (Experimental)
  Interventions: Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Bintrafusp alfa — Participants who are continuing treatment with bintrafusp alfa and were previously assigned to a bintrafusp alfa dose based on body weight which is (i.e.) milligrams per kilogram (mg/kg) dose in a parent protocol, will receive an intravenous infusion of bintrafusp alfa at the dose specified based upon the participant's parent protocol once every 2 week or, 2400 mg once every 3 weeks. Participants who are entering the rollover study after discontinuation of treatment in a parent study will receive bintrafusp alfa at a dose of either 1200 or 2400 mg once every 2 weeks or 2400 mg once every 3 weeks until confirmed disease progression, death, unacceptable toxicity or study withdrawal.
  Other Names: M7824

SUMMARY:
This study is designed to provide continuous access to treatment with bintrafusp alfa for eligible participants from ongoing bintrafusp alfa parent studies (NCT02517398, NCT02699515, NCT04246489, NCT03840915, NCT03631706, NCT04551950, NCT03833661 and NCT04066491) and to collect long-term safety and efficacy data.

Study Duration: All participants in this rollover study will be treated with bintrafusp alfa until meeting defined criteria in the protocol for discontinuation, until study intervention is commercially accessible and provisioned via marketed product, or until end of study.

The study also includes a 5 years survival follow-up after last dose of the study treatment.

Treatment Duration: Treatment under the rollover protocol according to the interval and dosing schedule in the parent protocol until discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are currently enrolled in an eligible bintrafusp alfa parent study where the primary/main analysis has been completed or after discontinuation of study before primary/main analysis has been completed or after discontinuation of study before primary/main analysis has been completed
* Participants who are currently on active bintrafusp alfa treatment alone as a monotherapy or following discontinuation of other combination treatment agents in the parent study and without treatment interruption at the time of rollover study enrollment
* Participants who experienced a confirmed complete response (CR), partial response (PR), or stable disease (SD) in an eligible parent study, discontinued bintrafusp alfa treatment according to the parent study protocol, and subsequently developed disease progression and are willing to re-start bintrafusp alfa treatment deemed potentially beneficial by the participants' physicians
* Participants who are.discontinued from bintrafusp alfa treatment in an eligible parent study due to an adverse events (AEs) that was subsequently well controlled or completely resolved after stopping therapy, provided that the parent study protocol permits reinitiation of bintrafusp alfa if a participant discontinued treatment due to toxicity and these participants are willing to re-start bintrafusp alfa treatment deemed potentially beneficial by the participants' physicians. Participants who have had AEs requiring permanent treatment discontinuation, like certain immune-related adverse events (irAEs) or certain bleeding events are excluded from participation in this Rollover study
* Participants with only SD at the time of discontinuation, the Investigator should confirm that no other reasonable treatment options are available
* Participants who have completed End of treatment (EoT) assessment of a parent study
* The investigator confirms that each participant agrees to use appropriate contraception and barriers, if applicable. The contraception, barrier, and pregnancy testing requirements are below:
* For female participants of childbearing potential or for male participants who have female partners of childbearing potential, the following applies:
* Participants on active treatment must agree to continue to use highly effective contraception for both male and female participants if the risk of conception exists thus, women of childbearing potential and men must agree to use highly effective contraception as stipulated in national or local guidelines
* Highly effective contraception must be used 28 days prior to the first study intervention administration, for the duration of study intervention, and at least for 2 months (for female participants) or 4 months (for male participants) after stopping study intervention
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the treating physician should be informed immediately

Exclusion Criteria:

* Participants who are pregnant or currently in lactation
* Participants with known hypersensitivity to any of the study intervention ingredients.
* Participants reinitiating treatment with bintrafusp alfa at study entry: have received any systemic anticancer therapies/treatments since discontinuing bintrafusp alfa treatment.
* Participants who has withdrawn consent from the parent study for any reason
* Any other reason that, in the opinion of the Investigator, precludes the participant from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (21):
- United States (2):
  - The Center for Cancer and Blood Disorders a Division of American Oncology Partners of Maryland, P.A., Bethesda, Maryland
  - NIH National Institutes of Health/GMB LTIB, Bethesda, Maryland
- Centre Hospitalier de l'Ardenne - PARENT, Libramont, Belgium
- Harbin Medical University Cancer Hospital, Harbin, China
- Universitaetsklinikum Carl Gustav Carus TU Dresden - Medizinische Klinik I, Dresden, Germany
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Lazio, Italy
- Japan (3):
  - National Cancer Center Hospital, Chūōku
  - Saitama Medical University International Medical Center, Hidaka-shi
  - National Cancer Center Hospital East, Kashiwa-shi
- BHI of Omsk region "Clinical Oncology Dispensary" - PARENT, Omsk, Russia
- South Korea (4):
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (3):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal - Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia - Servicio de Hematologia y Oncologia Medica, Valencia
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Chang Gung Memorial Hospital,Linkou, Taoyuan
- Adana City Hospital - Parent Account, Adana, Turkey (Türkiye)
- Communal Enterprise Volyn Regional Medical Center of Oncology of Volyn Regional Council - Department of Oncochemotherapy, Lutsk, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0054
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Biliary Tract Cancer: Participants with biliary tract cancer, who were continuing treatment with bintrafusp alfa and were previously assigned to a bintrafusp alfa dose based on body weight (i.e., milligrams per kilogram (mg/kg) dose) in a parent protocol (NCT02517398, NCT02699515, NCT04246489, NCT03840915, NCT03631706, NCT04551950, NCT03833661, and NCT04066491), received an intravenous infusion of bintrafusp alfa at the dose specified based upon the participant's parent protocol once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal. Participants who entered the rollover study after discontinuation of treatment in a parent study received bintrafusp alfa at a dose of either 1200 or 2400 mg once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal.
- Non-small Cell Lung Cancer: Participants with Non small cell lung cancer, who were continuing treatment with bintrafusp alfa and were previously assigned to a bintrafusp alfa dose based on body weight i.e., mg/kg dose in a parent protocol (NCT02517398, NCT02699515, NCT04246489, NCT03840915, NCT03631706, NCT04551950, NCT03833661, and NCT04066491), received an intravenous infusion of bintrafusp alfa at the dose specified based upon the participant's parent protocol once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal. Participants who entered the rollover study after discontinuation of treatment in a parent study received bintrafusp alfa at a dose of either 1200 or 2400 mg once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal.
- Cervical Cancer: Participants with cervical cancer, who were continuing treatment with bintrafusp alfa and were previously assigned to a bintrafusp alfa dose based on body weight i.e., mg/kg dose in a parent protocol (NCT02517398, NCT02699515, NCT04246489, NCT03840915, NCT03631706, NCT04551950, NCT03833661, and NCT04066491), received an intravenous infusion of bintrafusp alfa at the dose specified based upon the participant's parent protocol once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal. Participants who entered the rollover study after discontinuation of treatment in a parent study received bintrafusp alfa at a dose of either 1200 or 2400 mg once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal.
- Other (Colorectal Cancer, Glioblastoma, Melanoma): Participants with Other (Colorectal cancer, Glioblastoma, Melanoma) who were continuing treatment with bintrafusp alfa and were previously assigned to a bintrafusp alfa dose based on body weight i.e., mg/kg dose in a parent protocol (NCT02517398, NCT02699515, NCT04246489, NCT03840915, NCT03631706, NCT04551950, NCT03833661, and NCT04066491), received an intravenous infusion of bintrafusp alfa at the dose specified based upon the participant's parent protocol once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal. Participants who entered the rollover study after discontinuation of treatment in a parent study received bintrafusp alfa at a dose of either 1200 or 2400 mg once every 2 weeks or 2400 mg once every 3 weeks until disease progression, death, unacceptable toxicity, or study withdrawal.
Period: Overall Study
Arm/Group | Biliary Tract Cancer | Non-small Cell Lung Cancer | Cervical Cancer | Other (Colorectal Cancer, Glioblastoma, Melanoma)
Started | 10 | 5 | 3 | 4
Completed | 4 | 3 | 2 | 1
Not Completed | 6 | 2 | 1 | 3
Not completed — Death | 1 | 2 | 1 | 2
Not completed — End Of Study Due To Suspension Of Drug Supply | 2 | 0 | 0 | 0
Not completed — Stop By Sponsor | 2 | 0 | 0 | 1
Not completed — Poor protocol compliance led to sponsor-requested study withdrawal | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biliary Tract Cancer | Non-small Cell Lung Cancer | Cervical Cancer | Other (Colorectal Cancer, Glioblastoma, Melanoma) | Total
Number analyzed (Participants) | 10 | 5 | 3 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (10.3) | 63 (7.4) | 48 (14.4) | 52 (16.9) | 57 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 1 | 9
  Male | 7 | 3 | 0 | 3 | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Unknown or Not Reported | 10 | 5 | 3 | 4 | 22
  Race-Asian | 10 | 1 | 2 | 1 | 14
  Race-Black or African American | 0 | 1 | 0 | 0 | 1
  Race-White | 0 | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Related AEs (TRAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. TEAEs were defined as AEs emerging or worsening after start of treatment until 30 days after end of treatment. TRAE was defined as any AE considered as related to study treatment.
Time Frame: Baseline in parent study (NCT02517398, NCT02699515, NCT04246489, NCT03840915, NCT03631706, NCT04551950, NCT03833661 and NCT04066491) upto end of current rollover study (approximately assessed upto a maximum of 9 years, 6 months, 22 days)
Population: Safety analysis set included all participants who received at least one dose of study intervention in the Rollover study.
Measure: Count of Participants; unit: Participants
Arm/Group | Biliary Tract Cancer | Non-small Cell Lung Cancer | Cervical Cancer | Other (Colorectal Cancer, Glioblastoma, Melanoma)
Number analyzed (Participants) | 10 | 5 | 3 | 4
Participants
  TEAEs | 10 | 5 | 3 | 4
  TRAEs | 10 | 5 | 3 | 4

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from study day 1 in parent study to the date of death due to any cause. The overall survival was analyzed by using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS) included all participants who received at least one dose of study intervention in the Rollover study.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Biliary Tract Cancer | Non-small Cell Lung Cancer | Cervical Cancer | Other (Colorectal Cancer, Glioblastoma, Melanoma)
Number analyzed (Participants) | 10 | 5 | 3 | 4
months | NA [NA to NA] — Median overall survival and the upper and lower limits of the 90% confidence interval (CI) were not estimable due to an insufficient number of events. | NA [NA to NA] — Median overall survival and the upper and lower limits of the 90% CI were not estimable due to an insufficient number of events. | NA [NA to NA] — Median overall survival and the upper and lower limits of the 90% CI were not estimable due to an insufficient number of events. | NA [NA to NA] — Median overall survival and the upper and lower limits of the 90% CI were not estimable due to an insufficient number of events.

ADVERSE EVENTS:
Time Frame: From the first dose of study intervention in the Rollover study to the last administration of study intervention + 30 days (approximately 39 months and 21 days)
Arm/Group | Biliary Tract Cancer | Non-small Cell Lung Cancer | Cervical Cancer | Other (Colorectal Cancer, Glioblastoma, Melanoma)
All-Cause Mortality (participants affected / at risk) | 1/10 | 2/5 | 1/3 | 2/4
Serious Adverse Events (participants affected / at risk) | 3/10 | 4/5 | 1/3 | 2/4
Other Adverse Events (participants affected / at risk) | 8/10 | 3/5 | 3/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biliary Tract Cancer (N=10) | Non-small Cell Lung Cancer (N=5) | Cervical Cancer (N=3) | Other (Colorectal Cancer, Glioblastoma, Melanoma) (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biliary Tract Cancer (N=10) | Non-small Cell Lung Cancer (N=5) | Cervical Cancer (N=3) | Other (Colorectal Cancer, Glioblastoma, Melanoma) (N=4)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (18) | 1 (1) | 0 (0)
Ear swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Asthenia (General disorders) | 1 (2) | 2 (14) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (4) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (10) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05061823/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT05061823/SAP_001.pdf